CLINICAL TRIAL: NCT00985530
Title: A Phase I Trial of Tamibarotene and Arsenic Trioxide for the Treatment of Relapsed Acute Promyelocytic Leukemia
Brief Title: Tamibarotene and Arsenic Trioxide for Relapsed Acute Promyelocytic Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Supporting agency withdrew funding for study.
Sponsor: Northwestern University (Other)
Collaborators: CytRx (Industry); Cephalon (Industry)
Responsible Party: Principal Investigator, Jessica Altman, Jessica Altman, MD, Northwestern University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 08H9; NCI-2010-01852 (Other: NCI CTRP#); STU00012159 (Other: Northwestern University IRB#)
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Acute Promyelocytic Leukemia
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — tamibarotene; Arsenic Trioxide

ARMS (1):
- Arm 1 (Experimental): Tamibarotene + Arsenic Trioxide
  Interventions: Drug: Tamibarotene; Drug: Arsenic trioxide

INTERVENTIONS:
Drug: Tamibarotene — Self-administered tablets BID (approximately one hour after breakfast & dinner) during each 6 week cycle
Drug: Arsenic trioxide — Administered intravenously Monday thru Friday at 0.15 mg/kg - 30 doses per cycle.

SUMMARY:
Subjects have acute promyelocytic leukemia (APL) that has come back (relapsed) after initial treatment or has not gone away with initial therapy. This research study involves testing an investigational drug called Tamibarotene in combination with standard treatment for relapsed APL called arsenic trioxide. Tamibarotene has been approved in Japan to treat patients with relapsed APL since April 2005. Tamibarotene is in the same family of drugs as all-trans retinoic acid (ATRA), a medication that subjects received previously in their treatment. ATRA and tamibarotene both cause the APL cells to differentiate (or become) normal non-leukemia cells. Laboratory studies of tamibarotene have shown to be effective in APL. The purpose of this study is to determine if tamibarotene in combination with arsenic trioxide is safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* Must have diagnosis of relapsed APL
* Must have completed any prior cancer treatment at least 6 months prior to study
* Must have had prior treatment that included ATRA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To determine the safety and feasibility of combining tamibarotene and arsenic (ATO) for the treatment of patients with relapsed APL. | Once the MTD has been reached.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States